CLINICAL TRIAL: NCT06318117
Title: Observational Study on the Use of Infant Formulas Based on Rice Protein Hydrolysate in Real Life Conditions
Brief Title: Reason for Prescribing Rice Infant Formula
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Other Study IDs: 3398-1
Record Dates: First submitted 2024-03-06; First posted 2024-03-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Infant Formula
Keywords: Rice Formula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rice infant formula started before age of 6 months: After inclusion (V1), infants will return for a V2 visit at 12 months (± 30 days) of age (according to the child's regular appointment calendar). No visit is imposed by the protocol.
  Anthropometric data from visits to the pediatrician carried out between V1 and V2 will be collected from medical records, as well as the date of cessation of RIF, if applicable.
  Retrospective data will be collected from medical files (anthropometric data, medical and feeding history) and from parents' and investigator's recall.
  Interventions: Other: Rice infant formula
- Rice infant formula started after age of 6 months: After inclusion (V1), infants will return for a V2 visit at 12 months (± 30 days) of age (according to the child's regular appointment calendar). No visit is imposed by the protocol.
  Anthropometric data from visits to the pediatrician carried out between V1 and V2 will be collected from medical records, as well as the date of cessation of RIF, if applicable.
  Retrospective data will be collected from medical files (anthropometric data, medical and feeding history) and from parents' and investigator's recall.
  Interventions: Other: Rice infant formula

INTERVENTIONS:
Other: Rice infant formula — Any commercially available rice infant formula whom the pediatrician has previously deemed, or is deeming it useful to consume.

SUMMARY:
The main purpose of this study is to describe the pattern of RIF consumption in real life conditions, whatever the reasons of initiation and the chosen formula. The main objective is to study the reasons for prescribing a RIF during the first year of life, as per the pediatrician. Consumption started before 6 months of age, when milk and infantile formulas predominates in the baby's feeding, is of particular interest.

DETAILED DESCRIPTION:
The main purpose of this study is to describe the pattern of RIF consumption in real life conditions, whatever the reasons of initiation and the chosen formula. The main objective is to study the reasons for prescribing a RIF during the first year of life, as per the pediatrician. Consumption started before 6 months of age, when milk and infantile formulas predominates in the baby's feeding, is of particular interest. Secondary objectives are to describe the modalities of feeding before, during and after consuming the RIF, to describe the growth of children who have consumed a RIF for at least 1 month, on the basis of anthropometric data collected during the first year of life. As a second intention, this study also aims to monitor the evolution of child's digestive and allergic symptoms, if any, and the sociodemographic characteristics of the infant's family.

ELIGIBILITY:
Inclusion Criteria:

* Child aged between 6 and 36 months,
* Child who has already consumed a RIF for at least one month, or still consuming a RIF, or who will benefit from taking a RIF, according to the pediatrician,
* Legal representatives (parents/guardians) deemed capable of following the requirements of the protocol and have given their consent orally.

Exclusion Criteria:

* Child with a clinically relevant and significant abnormality in the medical history or on physical examination;
* Child who has been hospitalized in a neonatology unit (due to prematurity, malformation or neonatal pathology), or born with a low birth weight (≤ 2,500 g);
* For children not diversified at the time of starting RIF: mixed feeding with RIF and breast milk and/or infant formula based on cow's milk;
* Child born to minor parent(s);
* Infant or infant's family unable to comply with study protocol or procedures, in the judgment of the investigator;
* Participation in any other clinical trial prior to inclusion;
* Refusal of the Parents / legal representatives of the child, or who do not master the French language well enough to understand the information letter.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 infants will be recruited for this study, according to the following inclusion and non-inclusion criteria, including at least 60 infants who started the RIF before the age of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire - reason for prescribing a RIF during the 1st year of life. | 1 to 7 months
  The main objective is to describe the main reason for prescribing a RIF by the pediatrician during the 1st year of life.

SECONDARY OUTCOMES:
Questionnaire - Reason for prescribing a RIF in first 6 months of life | up to 365 days of age
  o describe the main reason for prescribing a RIF by the pediatrician during the 1st 6 months of life.
Questionnaire - Diet characteristics | up to 365 days of age
  To describe the conditions of RIF consumption during the follow-up, and the other main characteristics of the diet.
Growth z-scores body mass index (BMI)-for-age | up to 365 days of age
  body mass index (BMI)-for-age
Growth z-score | up to 365 days of age
  Weight-for-age z-score
Growth z-score | up to 365 days of age
  Length/Height-for-age z-score
Growth z-score | up to 365 days of age
  Weight-for-length/height z-score
Growth z-score | up to 365 days of age
  Head circumference-for-age z-score
Questionnaire - Evolution of digestive and allergic symptoms | up to 365 days of age
  To describe the evolution of digestive and allergic symptoms during follow-up.
Socio-demographic characteristics | up to 365 days of age
  To describe the socio-demographic characteristics of the infants' families

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Piloquet, MD, Principal Investigator — CHU Nantes Children's chronic disease service
Locations (17):
- France (17):
  - Centre Hospitalier d'Auxerre - Neonatology and pediatric emergency department, Auxerre, Auxerre
  - Dr Christine REGIMBART - Private Practice, Bécon-les-Granits, Becon-les-Granits
  - Scm Les Pediatrices Du Pic St Loup, Saint-Clément, DE Riviere
  - Dr. Anne Sengier - Private Practice, Le Havre, LE Havre
  - Centre Hospitalier de Montauban - Pediatric Department, Montauban, Montauban
  - Centre Hospitalier Universitaire de Nantes - Pediatric emergency department, Nantes, Nantes
  - Hôpital NOVO - Pediatric department, Pontoise, Pontoise
  - Dr Marta Nowak-Mohamed - Private Practice, Vichy, Vichy
  - Dr Frederic Couttenier Private Practice, Attiches
  - Elise Foy-Foulkes Private Practice, Boulogne-Billancourt
  - Dr. Anne Cheve Private Practice, Brest
  - Dr. Sandra Brancato Private Practice, Brignon
  - Dr. Karim Abada Private Practice, Foix
  - Dr. Nellie Houeto Private Practice, Hyères
  - Dr. Amandine Blasquez Private Practice, Libourne
  - Dr. Marc Sznajder Private Practice, Paris
  - Dr. Piotr Gembara Private Practice, Vichy

IPD SHARING:
Plan to Share IPD: No